CLINICAL TRIAL: NCT05865821
Title: Protocol Effect of Negative Pressure Drain to Reducing Surgical Site Infection in Clean-contaminated and Contaminated Surgical Wound of Abdominal Surgery
Brief Title: Protocol Effect of Negative Pressure Drain to Reducing Surgical Site Infection in Surgical Wound of Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MURA2023/168
Record Dates: First submitted 2023-05-04; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Surgical Site Infection
Keywords: abdominal surgery, surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Negative pressure drainage is a drainage catheter which is placed in subcutaneous surgical wound for draining fluid such as hematoma, seroma, and pus. In this study the drainage the catheter will be placed in the wound for 5 days and/or removed if fluid content is less than 20 ml per day. Jackson-Pratt catheter is used in this study because it is cheap and widespread in all hospitals. The drainage catheter is placed after completion of surgery and before skin closure.
Who Masked: Investigator
Masking Description: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative pressure drainage (Active Comparator): Negative pressure drainage is a drainage catheter which is placed in subcutaneous surgical wound for draining fluid such as hematoma, seroma, and pus. In this study the drainage the catheter will be placed in the wound for 5 days and/or removed if fluid content is less than 20 ml per day. Jackson-Pratt or Redivac catheter is used in this study because it is cheap and widespread in all hospitals. The drainage catheter is placed after completion of surgery and before skin closure.
  Interventions: Procedure: Negative pressure drainage
- No pressure drain (Other): no drainage catheter in subcutaneous surgical wound
  Interventions: Other: No pressure drain

INTERVENTIONS:
Procedure: Negative pressure drainage — Negative pressure drainage is a drainage catheter which is placed in subcutaneous surgical wound for draining fluid such as hematoma, seroma, and pus. In this study the drainage the catheter will be placed in the wound for 5 days and/or removed if fluid content is less than 20 ml per day. Jackson-Pratt catheter or Redivac is used in this study because it is cheap and widespread in all hospitals. The drainage catheter is placed after completion of surgery and before skin closure
  Arms: Negative pressure drainage
Other: No pressure drain — Negative pressure drainage is a drainage catheter which is placed in subcutaneous surgical wound for draining fluid such as hematoma, seroma, and pus. In this study the drainage the catheter will be placed in the wound for 5 days and/or removed if fluid content is less than 20 ml per day. Jackson-Pratt catheter or Redivac is used in this study because it is cheap and widespread in all hospitals. The drainage catheter is placed after completion of surgery and before skin closure
  Arms: No pressure drain

SUMMARY:
Surgical site infection (SSI) is one of main complication in surgery. It usually occurs within 30 days post operation. The superficial SSI is an infection of skin and subcutaneous layer, clinically presented by pus oozing. Furthermore, seroma hematoma and wound dehiscence are also clinical signs of superficial SSI.

Nowadays, there are studies which report methods reducing SSI by placing negative pressure drain within surgical wound. It can reduce serum in subcutaneous layer which is found in every surgical wound, especially in clean-contaminated and contaminated wound. Many studies show that placing negative pressure drainage within a surgical wound can reduce superficial SSI and decrease hospital length of stay by comparing with the control group.

The objective in this study to compare the rate of SSI of clean-contaminated and contaminated surgical wounds between the patients whose wounds are placed with negative pressure drainage and patients who were not placed with negative pressure drainage.

DETAILED DESCRIPTION:
This study is a randomized controlled trial, double-blinded and performs in the patient who underwent intra-abdominal surgery. the investigators collect the data at the department of surgery, Ramathibodi hospital. This study randomized the volunteer patient into 2 groups as follow: the patient with placing negative pressure drainage within the surgical wound and the patient without placing negative pressure drainage.

* Randomization To minimize the study bias, the investigators random patient into two groups by the unassociated personnel opens an enclosed envelope after the surgical procedure is completely performed and before the beginning of closing the skin layer.
* Blind process This study does not conceal information about surgical technique and drain placing method. However, the investigators have controlled various surgical procedures to reduce inequality in assessment and bias.
* Negative pressure drainage is a drainage catheter which is placed in surgical wound for draining fluid such as hematoma, seroma, and pus. In this study the drainage the catheter will be placed in the wound for 5 days and/or removed if fluid content is less than 20 ml per day. Jackson-Pratt or Redivac catheter is used in this study because it is cheap and widespread in all hospitals. The drainage catheter is placed after completion of surgery and before skin closure.
* Surgical site infection (SSI) is infection at surgical wound which happens within 30 days post operatively and in this study will use in term of superficial SSI (pus oozing, cellulitis and wound culture positive) If patients have SSI, the investigators remove the drain from the patients (intervention group) and may total stitch off suture then wet dressing combine with antibiotic.

the investigators evaluate and collect data by physical examination at post operation day 3, day 5,day 7 and the day that patient is discharged from hospital. Then investigators follow up the patients at 14 days and 30 days after discharged from hospital.The complication of SSI is seroma, hematoma and wound dehiscence.

* Seroma is the retention of clear fluid in the cavity of the body such as a surgical wound. Typical clinical presentation is fluid oozing from the wound.
* Hematoma is the retention of bloody fluid in the cavity of the body such as a surgical wound. It can be infected which is possible to prevent by stop bleeding intraoperatively and evaluate surgical wound every day.
* Wound dehiscence is partial or total separation of previously approximated wound edges, due to failure of proper wound healing.

In patient case with infected wound and the investigators give antibiotics along with dressing, but does not stitch off suture, we do not include as SSI in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing intra-abdominal surgery on the upper and lower gastrointestinal tract, pancreas and biliary tract.
* Aged 18 years or older
* Be in good health and full of consciousness.
* Willing to participate in the research study project by signing

Exclusion Criteria:

* Patients with thrombocytopenia thrombocytopenia or coagulation disorder
* The study participant refuses or withdraws from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-03-06 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of SSI | post operation day 3
  To compare the rate of SSI of clean-contaminated and contaminated surgical wounds between the patients whose wounds are placed with negative pressure drainage and patients who were not placed with negative pressure drainage
Rate of SSI | post operation day 5
  To compare the rate of SSI of clean-contaminated and contaminated surgical wounds between the patients whose wounds are placed with negative pressure drainage and patients who were not placed with negative pressure drainage
Rate of SSI | post operation day 7
  To compare the rate of SSI of clean-contaminated and contaminated surgical wounds between the patients whose wounds are placed with negative pressure drainage and patients who were not placed with negative pressure drainage
Rate of SSI | post operation day 14
  To compare the rate of SSI of clean-contaminated and contaminated surgical wounds between the patients whose wounds are placed with negative pressure drainage and patients who were not placed with negative pressure drainage

SECONDARY OUTCOMES:
Length of hospital stay | day 3
  amount of days that the patient stay in hospital since admission date until discharged from the hospital.
Length of hospital stay | day 5
  amount of days that the patient stay in hospital since admission date until discharged from the hospital.
Length of hospital stay | day 7
  amount of days that the patient stay in hospital since admission date until discharged from the hospital.
Length of hospital stay | day 14
  amount of days that the patient stay in hospital since admission date until discharged from the hospital.
Score of Quality of life | day 7
  Quality of life is patient's physical health and mental health. We collect this data by 36-Item Short Form Survey Instrument (SF-36) survey at the 7th day and 14th day after being discharged from the hospital
Score of Quality of life | day 14
  Quality of life is patient's physical health and mental health. We collect this data by 36-Item Short Form Survey Instrument (SF-36) survey at the 7th day and 14th day after being discharged from the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Chairat Supsamutchai, MD, Study Chair — Ramahibodi hospital, Mahidol University; Ninnat Fongsupa, MD, Principal Investigator — Ramahibodi hospital, Mahidol University; Napaphat Poprom, Ph.D, Study Director — Ramahibodi hospital, Mahidol University
Locations (1):
- Chairat Supsamutchai, Bangkok, Bankok, Thailand

IPD SHARING:
Plan to Share IPD: No